CLINICAL TRIAL: NCT03121677
Title: Pilot Study of a Personalized Tumor Vaccine Strategy and PD-1 Blockade in Patients With Follicular Lymphoma
Brief Title: Personalized Tumor Vaccine Strategy and PD-1 Blockade in Patients With Follicular Lymphoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Vaccine manufacturing has been suspended
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201804151
Record Dates: First submitted 2017-04-17; First posted 2017-04-20 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Follicular Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular | interventions — poly ICLC; Nivolumab; Leukapheresis; Rituximab; Biopsy

STUDY DESIGN:
Intervention Model Description: For the first three patients treated on study therapy, treatment of each subsequent patient will not be allowed until the prior patient has completed Cycle 1. If no unexpected adverse events attributed to the combination therapy are observed, after the third patient completes Cycle 1, treatment initiation may occur without restrictions for the remaining patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Nivolumab/Poly-ICLC/Vaccine/+/- Rituximab (Experimental): * All cycles are 4 weeks (wks), with nivolumab every 2 wks during Cycles 1-6 & every 4 wks during Cycles 7-12 & vaccine on Cycle 1 Days 1, 4, 8, 15; Cycle 2 Day 1; and then on Day 1 of Cycles 4, 6, 8, 10, 12
  * After 2 cycles, restaging will be performed, & patients with CR, PR, or SD will continue on nivolumab + vaccine. Patients with evidence of PD may initiate anti-CD20 mAb therapy (drug to be determined by the treating physician) weekly for 4 wks during Cycle 3, followed by a dose on Day 1 of every other cycle (Cycles 6, 8, 10, and 12).
  * After 6 cycles, restaging will be performed again, and patients with CR, PR, or SD will continue nivolumab + vaccine. Patients with PD at that time point (but not treated with anti-CD20 mAb therapy thus far on this protocol) will initiate anti-CD20 mAb (drug to be determined by the treating physician) therapy weekly for 4 wks during Cycle 7, followed by a dose Day 1 of Cycles 10 & 12 & 2 additional doses 8 wks apart.
  Interventions: Biological: Personalized tumor vaccine; Drug: Poly ICLC; Biological: Nivolumab; Procedure: Peripheral blood draws; Procedure: Leukapheresis; Biological: Rituximab; Procedure: Biopsy

INTERVENTIONS:
Biological: Personalized tumor vaccine — * Cycle 12 vaccine administration is optional
  * The peptides comprising the vaccine are reconstituted in up to 4 pools with 5 peptides per pool (A, B, C, and D) . At each vaccination time point, each of the up to four pools will be administered to one of the four limbs (A - Right Arm, B - Left Arm, C - Right Leg, D - Left Leg) by subcutaneous injection.
Drug: Poly ICLC — -The personalized tumor vaccine will be co-administered with poly-ICLC.
  Other Names: poly-ICLC
Biological: Nivolumab — -Nivolumab will be administered at a dose of 240 mg intravenously
  Other Names: Opdivo
Procedure: Peripheral blood draws — -Time of biopsy, during the pre-treatment check (any time before cycle 1 day 1), Cycle 1 Day 15, Cycle 2 Day 1, Cycle 3 Day 1, Cycle 4 Day 1, Cycle 6 Day 1, Cycle 12 Day 1, Time of response, and Time of progression or relapse
Procedure: Leukapheresis — * Prior to the initiation of treatment and up to five days prior to treatment on cycle 6 day 1, patients will undergo apheresis according to standard institutional procedures for non-mobilized collection.
  * Peripheral blood leukocytes will be cryopreserved for later assessment for the presence of T-cells that recognize tumor specific mutant antigens and immunophenotype, and the presence of other lymphocytes or regulatory populations.
Biological: Rituximab — -Other anti-CD20 mAb treatment can be used
  Other Names: Rituxan
Procedure: Biopsy — -Biopsies on lymph node or extranodal site(s) are to be obtained at: screening (only after the patient is deemed eligible; during cycle 2 (after treatment on C2D15 and prior to treatment on C3D1); disease relapse or progression (if this occurs)

SUMMARY:
Follicular lymphoma (FL) has a number of effective standard of care therapies; however, FL is not currently considered curable. Therefore, designing well tolerated therapies without cumulative and long-term toxicity is critical. This is a pilot safety and feasibility study that combines a personalized tumor vaccine with nivolumab for the treatment of FL. Patients who demonstrate progression on this study may be treated with rituximab (or another monoclonal antibody against CD20) in addition to vaccine therapy with nivolumab at the discretion of treating physician if clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed follicular lymphoma, grade 1-3a
* Patients who have relapsed after at least 1 prior anti-lymphoma therapy that include anti-CD20 monoclonal antibody and an alkylator chemotherapy agent, or at least 2 prior anti-lymphoma therapies that include anti-CD20 monoclonal antibody, may be included
* Anti-CD20 mAb-naïve or anti CD20 mAb-sensitive (defined as progression of FL ≥ 6 months following prior anti-CD20 mAb containing therapy).
* Presence of measurable disease according to the 2014 Lugano Classification
* Disease course appropriate for therapy initiation approximately 4-5 months from enrollment per treating physician.
* Tumor site amenable to a) excisional biopsy or b) approximately 12 core biopsies from lymph node or extranodal site(s) or other site of lymphoma or c) other surgical procedure to provide adequate lymphoma sample for TSMA sequencing and screening.
* At least 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1
* Normal bone marrow and organ function as defined below:

  * Absolute neutrophil count ≥ 1,000/mcl
  * Platelets ≥ 100,000/mcl
  * Total bilirubin ≤ 1.5 x ULN
  * AST, ALT ≤ 3.0 x ULN
  * Creatinine clearance ≥ 50 mL/min (calculated by the Cockcroft-Gault or via 24-hour urine collection)
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Known current or previous histologic transformation from indolent non-Hodgkin lymphoma to diffuse large B-cell lymphoma or other aggressive lymphoma histology.
* Any anti-lymphoma treatment within 6 months' treatment initiation.
* Prior therapy with anti-PD-1, PD-L1, or PD-L2 agent.
* Diagnosis of a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Live vaccine within 30 days prior to treatment initiation.
* Prior organ allograft or allogeneic transplantation.
* Known central nervous system (CNS) involvement with lymphoma.
* Tested positive for hepatitis B surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or chronic infection.
* Known history of HIV or AIDS.
* History of concurrent malignancy requiring active therapy or prior history of another malignancy within 5 years
* Active, known, or suspected autoimmune disease. Subjects are permitted to enroll if they have vitiligo, type 1 diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in absence of an external trigger.
* Currently receiving any other investigational agents.
* A history of allergic reactions or significant toxicity attributed to compounds of similar chemical or biologic composition to anti-CD20 mAbs, anti-PD-1 mAbs, or TLR agonists.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* Women who are pregnant and/or breastfeeding. Women of childbearing potential must have a negative serum or urine pregnancy test within 24 hours prior to the start of nivolumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2023-08-07 (Actual)

PRIMARY OUTCOMES:
Feasibility and safety of vaccine in combination with nivolumab +/1 anti-CD20 monoclonal antibody therapy as measured by the number of participants whose personal vaccines can be manufactured and delivered without unacceptable toxicity | Through 6 months following the first treatment of the last patient enrolled (approximately 54 months)
  -Unacceptable toxicity will be described as inability to receive further therapy due to toxicities of therapy as defined by NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 or the occurrence of other toxicities deemed to be at sufficiently high risk to patients by the principal investigator

SECONDARY OUTCOMES:
Overall response rate (ORR) | Through 5 years after completion of treatment (approximately 111 months)
  * ORR = number of participants with complete response + number of participants with partial response
  * Overall response rates will be compared between participants who received anti-CD20 mAb treatment (rituximab) versus those participants who did not receive anti-CD20 mAb treatment
Complete response (CR) rate | Through 5 years after completion of treatment (approximately 111 months)
  * CR rates will be compared between participants who received anti-CD20 mAb treatment (rituximab) versus those participants who did not receive anti-CD20 mAb treatment
  * CR:
    * Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
    * London Deauville score of 1 and 2 in lymph nodes and extra lymphatic sites is considered to represent complete metabolic response. A London Deauville score 3 in the post treatment PET scan may be considered to represent complete metabolic response especially if it is not higher than the surrounding normal physiologic uptake.
    * No evidence of FDG avid disease in the bone marrow
    * No new lesions
    * If the bone marrow was involved by lymphoma before treatment, the infiltrate must have cleared on repeat bone marrow biopsy.
Duration of response | Through 5 years after completion of treatment (approximately 111 months)
  * Duration of responses will be compared between participants who received anti-CD20 mAb treatment (rituximab) versus those participants who did not receive anti-CD20 mAb treatment
  * Duration of response = time from first vaccine dose to first evidence of disease progression in participants with at least one response of CR, PR, or SD
Progression-free survival (PFS) | Through 5 years after completion of treatment (approximately 111 months)
  * PFS will be compared between participants who received anti-CD20 mAb treatment (rituximab) versus those participants who did not receive anti-CD20 mAb treatment
  * PFS: time from first CR, PR, or SD response to disease progression, death, or last follow-up
  * PD:
    * London Deauville score of 4 or 5 in individual target nodes/masses with an increase in intensity of uptake from the baseline and/or new FDG avid foci consistent with lymphoma at interim or end of treatment assessment
    * New FDG avid foci of extranodal disease consistent with lymphoma. If there is concern regarding the etiology of the new lesions, biopsy or interval scan may be considered.
    * New or recurrent FDG avid foci in the bone marrow
Overall survival (OS) | Through 5 years after completion of treatment (approximately 111 months)
  * OS will be compared between participants who received anti-CD20 mAb treatment (rituximab) versus those participants who did not receive anti-CD20 mAb treatment
  * OS: time from first vaccine dose to death or last follow-up
Partial response (PR) rate | Through 5 years after completion of treatment (approximately 111 months)
  * Partial response rates will be compared between participants who received anti-CD20 mAb treatment (rituximab) versus those participants who did not receive anti-CD20 mAb treatment
  * PR:
    * London Deauville score of 4 or 5 in lymph nodes and extra lymphatic sites with reduced uptake compared with the baseline and residual mass(es) of any size on interim scan
    * Residual bone marrow uptake higher than the uptake in the normal marrow but reduced when compared with baseline If there are persistent focal changes in the marrow in the context of a nodal response consideration should be given to further evaluation with MRI or biopsy or an interval scan
    * No new lesions

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Bartlett, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ramirez CA, Becker-Hapak M, Singhal K, Russler-Germain DA, Frenkel F, Barnell EK, McClain ED, Desai S, Schappe T, Onyeador OC, Kudryashova O, Belousov V, Bagaev A, Ocheredko E, Kiwala S, Hundal J, Skidmore ZL, Watkins MP, Mooney TB, Walker JR, Krysiak K, Gomez F, Fronick CC, Fulton RS, Schreiber RD, Mehta-Shah N, Cashen AF, Kahl BS, Ataullakhanov R, Bartlett NL, Griffith M, Griffith OL, Fehniger TA. Neoantigen landscape supports feasibility of personalized cancer vaccine for follicular lymphoma. Blood Adv. 2024 Aug 13;8(15):4035-4049. doi: 10.1182/bloodadvances.2022007792. PMID 38713894
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu